CLINICAL TRIAL: NCT05778474
Title: Mechanical Determinants of Upper Limbs Oscillation During Gait
Acronym: CLAPENDAS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 24C901_2019
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Poststroke/CVA Hemiparesis; Parkinson Disease; Cerebral Palsy; Amputation
Keywords: Walking; Upper limb oscillations; Treadmill; Center of Mass; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: At least 10 healthy participants aged from 18 to 60 years old with symmetric walking at visual analysis. Participants will be excluded if pregnant, if they present with pharmacologic therapies which could affect balance and walking, and if they suffered from (or presently present with) orthopedic or neurologic conditions potentially impairing walking.
  Interventions: Other: Healthy subjects
- Pathologic group: At least 15 participants with various orthopaedic or neurologic conditions (for example, post-stroke hemiparesis, Parkinson's disease, multiple sclerosis, unilateral amputation, surgical orthopedic interventions) will be enrolled. Participants will present a unilateral motor impairment, not preventing passive oscillation of the upper limbs.
  Interventions: Other: Pathologic group

INTERVENTIONS:
Other: Healthy subjects — Participants' ground spontaneous speed overground will be tested by means of the 10-meter walking test. Participants will be tested for their foot dominance by means of the Waterloo footedness questionnaire-revised. Participants will walk on a treadmill mounted on force sensors. The test sequence will be the following:
  1. Familiarization. Participants will walk on the treadmill with the belt running at increasing velocities up to their spontaneous walking velocity . Speed will be increased of 0.2 m s-1 every 30 s. A brief pause of around 1 minute will follow.
  2. Walking. Participants will walk at 0.4 m s-1 and 1.2 m s-1 for at least 30 seconds.
  3. Walking with a rigid ankle-foot orthosis. Participants will walk at 0.4 m s-1 and 1.2 m s-1 for at least 30 seconds with an ankle-foot orthosis on the dominant lower limb.
  Participants will repeat the last point (n°3) with the ankle-foot orthosis on the non-dominant lower limb. A 3-min pause will follow each section.
  Groups: Healthy participants
Other: Pathologic group — Participants will walk on a treadmill mounted on force sensors. They will walk freely, under tight supervision, but without hanging to any support. The test sequence will be the following:
  4. Familiarization. Participants will walk on the treadmill with the belt running at increasing velocities up to their spontaneous walking velocity . Speed will be increased of 0.1 m s-1 every 30 s. A brief pause of around 1 minute will follow.
  5. Walking. Participants will walk at 0.4 m s-1 for at least 30 seconds. Participants will be informed a few seconds before the changes in belts' velocities with a verbal warning.
  Groups: Pathologic group

SUMMARY:
It is unclear why humans typically swing their arms during gait. To date, the debate on how to arm swing comes about (i.e. whether it is caused by accelerations of the shoulder girdle or muscular activity) is still going on. There needs to be consensus on whether the arm swing is actively controlled or merely passive and on why humans swing their arms during walking (i.e. what the purpose of arm swing is, if any). Suggested reasons include minimising energy consumption, optimising stability, and optimising neural control. Pathologies such as hemiplegia after stroke, Parkinson's disease, Cerebral Palsy, Spinal Cord Injury, and Multiple Sclerosis may directly affect arm swing during gait. Emerging evidence indicates that including arm movements in gait rehabilitation may be beneficial in restoring interlimb coordination and decreasing energy expenditure.

This project hypothesises that the arms swing, at least at low and intermediate walking speeds, reflects the body's Center of Mass (CoM) accelerations. Arm swing may thus depend mainly upon the system's intrinsic mechanical properties (e.g., gravity and inertia). In this perspective, the CoM is seen as moving relative to the upper limbs rather than the other way around. The contribution of major lower limb joints, in terms of power injected into the body motion, will be simultaneously explored.

The study aims to investigate the mechanism and functions of arm swinging during walking on a force treadmill. To simulate asymmetric walking, healthy subjects will be asked to walk with a toes-up orthosis to induce claudication and asymmetry in ankle power. In this way, it will be possible to highlight the correlation among arm swinging, ankle power, and the acceleration of the CoM in a 3D framework. In addition, subjects affected by unilateral motor impairments will be asked to walk on the force treadmill to test the experimental model and highlight significant differences in the kinematic parameters of the upper limbs.

The question of whether arm swing is actively controlled or merely passive and the relationship between arm swinging and the total mechanical energy of the CoM will be faced.

Asymmetric oscillations of the upper limb will be related to dynamic asymmetries of the COM motion, and of the motion of lower limbs. In addition, cause-effect relationships will be hypothesized. Finally, the dynamic correlates of upper limb oscillations will make the clinical observation an interpretable clinical sign applicable to rehabilitation medicine.

Results from the present study will also foster the identification of practical rehabilitation exercises on gait asymmetries in many human nervous diseases.

ELIGIBILITY:
Inclusion Criteria:

* presence of claudication (spatiotemporal asymmetry between subsequent steps), at visual inspection;
* unilateral motor impairments of one lower limb as a consequence of various pathologic conditions, such as (not not limited to): poststroke hemiparesis (ischemic or hemorrhagic), Parkinson's disease, multiple sclerosis, unilateral amputation with prosthetic correction, surgical orthopedic interventions;
* ability to walk for at least 100 meters without support; prostheses or orthoses admitted.
* ability to wittingly sign the informed consent form

Exclusion Criteria:

* drug therapy underway up to three months before recruitment, with impact on balance and gait;
* systemic pathologies or other sensory or neurological pathologies with impact on balance and gait;
* Mini Mental State (MMSE) score < 24/30;
* alterations in the passive mobility of upper limbs;
* painful syndrome which could alter the locomotion;
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be recruited in the proponent Unit on an outpatient basis, from a physiatric referral or from a local inpatient rehabilitation unit.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Ankle joint power | Day 1
  Joint kinematics will be recorded through an optoelectronic method as per the Davis anthropometric model. The 3D displacement of the markers will be captured using 10 near-infrared stroboscopic cameras. Joint power will be computed through the spatiotemporal synchronization of ground reaction force vectors and the joint centers of rotation. The sagittal plane will be only considered for the analysis. Joint power will be computed as the product of joint torque and joint rotation speed. Power will be defined as positive or generated when the joint moment and rotation speed shared the same directions (i. e., when agonist muscles are contracting while shortening), as negative or absorbed otherwise. Positive work will be computed as the integral of the generated (positive) power over time.

SECONDARY OUTCOMES:
Spatio parameter | Day 1
  Step length: the sagittal distance between the markers put on the lateral malleolus of the posterior and anterior feet at the ground strike of the anterior foot.
  The Step length is measured in meters [m].
Shoulder and elbow joint angles on the sagittal plane | Day 1
  Shoulder flexion-extension angle, Elbow flexion-extension angle. Angle is measured in degrees (deg.)
Energy of the center of mass | Day 1
  The changes in kinetic energy due to the forward (Ekf), lateral (Ekl) and vertical (Ekv) velocity; the changes of gravitational potential energy (Ep); the changes of the mechanical energy due to the vertical motion, Ev = Ekv+Ep; the changes of the total mechanical energy (Etot = Ekf+Ekl +Ev). Amounts of energy are measured in Joule/Kg.

OTHER OUTCOMES:
Time parameters | Day 1
  Single Stance Time: for each lower limb, the time interval during which the limb determines vertical ground reactions equal to or exceeding 30 N.
  Double Stance Time: the time interval during which, under both lower limbs, vertical ground reactions equal or exceed 30 N.
  Time parameters are measured in seconds [s].
The trajectory of the center of mass | Day 1
  the trajectory of the centre of mass will be studied in the sagittal and frontal planes during the strides. will be measured in meters [m].

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Tesio, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rota V, Caronni A, Scarano S, Amadei M, Tesio L. Plantar flexors are the main engine of walking in healthy adults. Front Sports Act Living. 2025 Jul 8;7:1595065. doi: 10.3389/fspor.2025.1595065. eCollection 2025. PMID 40697531